CLINICAL TRIAL: NCT05405218
Title: Trial of Ultrasound Guided Carpal Tunnel Release Versus Traditional Open Release (TUTOR)
Acronym: TUTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonex Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90079-TP
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome; CTS; Carpal Tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carpal Tunnel Release with Ultrasound Guidance using the UltraGuideCTR device (Experimental)
  Interventions: Device: CTR with Ultrasound Guidance using the UltraGuideCTR device
- Mini Open Carpal Tunnel Release (mOCTR) (Active Comparator)
  Interventions: Procedure: mOCTR

INTERVENTIONS:
Device: CTR with Ultrasound Guidance using the UltraGuideCTR device — Carpal Tunnel Release with Ultrasound Guidance using UltraGuideCTR device
  Arms: Carpal Tunnel Release with Ultrasound Guidance using the UltraGuideCTR device
Procedure: mOCTR — Mini Open Carpal Tunnel Release
  Arms: Mini Open Carpal Tunnel Release (mOCTR)

SUMMARY:
Study to compare the safety and effectiveness of carpal tunnel release with ultrasound guidance (CTR-US) vs. mini-open carpal tunnel release (mOCTR) in patients with symptomatic carpal tunnel syndrome (CTS).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Clinical diagnosis of unilateral or bilateral idiopathic CTS
3. CTS-6 score >12 in target hand
4. Absence of carpal tunnel symptoms in the contralateral hand that interfere with normal daily activities or work at the time of consent and are not anticipated to interfere with return to activities or return to work within at least 3 months post-operatively
5. Median nerve cross-sectional area ≥10 mm2 in the proximal carpal tunnel region of the target hand measured by diagnostic ultrasound
6. Prior failure of one or more nonsurgical treatment options for the target hand (e.g., physical activity modification, bracing, splinting, corticosteroid injection)
7. Subject agrees to complete follow-up questionnaires over a 12-month period
8. Subject has a valid mobile phone number and email address to receive and answer follow-up questionnaires

Exclusion Criteria:

1. Prior surgery on the target wrist or hand with the exception of trigger finger that has clinically recovered
2. History of prior surgical CTR procedure in the target hand
3. History of prior surgical CTR in the contralateral hand within 3 months of enrollment or with persistent symptoms that interfere with normal daily activities or work at the time of consent
4. Corticosteroid injection in the target wrist or hand within 6 weeks of study procedure date
5. Presence of additional process in the target wrist or hand requiring additional intervention beyond carpal tunnel release (e.g. neurolysis, mass removal, tenosynovectomy)
6. Clinically significant degenerative arthritis of the upper limb (shoulder to hand) on the target side
7. Clinically significant inflammatory disease (including tenosynovitis) of the upper limb (shoulder to hand) on the target side
8. Clinically significant trauma or deformity of the upper limb (shoulder to hand) on the target side
9. Clinically significant vascular disease (including Raynaud's phenomenon) of the upper limb (shoulder to hand) on the target side
10. Clinically significant neurological disorder (including complex regional pain syndrome) of the upper limb (shoulder to hand) on the target side
11. Planned surgical or interventional procedure on the contralateral wrist or hand
12. Systemic inflammatory disease (e.g., rheumatoid arthritis, lupus)
13. Amyloidosis
14. Chronic renal insufficiency requiring dialysis
15. Diabetes not controlled by a stable dose of medication over the past three months
16. Uncontrolled thyroid disease
17. Pregnant or planning pregnancy in the next 12 months
18. Workers compensation subjects
19. Inability to provide a legally acceptable Informed Consent Form and/or comply with all follow-up requirements
20. Subject has other medical, social or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Eberlin, MD, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (12):
  - Sierra Orthopedic Institute, Sonora, California
  - Orthopedic Associates, Fort Walton Beach, Florida
  - Tri-State Orthopaedics, Evansville, Indiana
  - Indiana Hand to Shoulder, Indianapolis, Indiana
  - Kansas Orthopaedic Center, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Twin Cities Orthopedics, Plymouth, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - Midwest Orthopedic Group, Farmington, Missouri
  - Sano Orthopedics, Lee's Summit, Missouri
  - Washington University, St Louis, Missouri
  - ATX Orthopedics, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eberlin KR, Amis BP, Berkbigler TP, Dy CJ, Fischer MD, Gluck JL, Kaplan FTD, McDonald TJ, Miller LE, Palmer A, Perry PE, Walker ME, Watt JF. Multicenter randomized trial of carpal tunnel release with ultrasound guidance versus mini-open technique. Expert Rev Med Devices. 2023 Jul;20(7):597-605. doi: 10.1080/17434440.2023.2218548. Epub 2023 May 30. PMID 37254502
- [Derived] Eberlin KR, Dy CJ, Fischer MD, Gluck JL, Kaplan FTD, McDonald TJ, Miller LE, Palmer A, Walker ME, Watt JF. Trial of ultrasound guided carpal tunnel release versus traditional open release (TUTOR). Medicine (Baltimore). 2022 Oct 14;101(41):e30775. doi: 10.1097/MD.0000000000030775. PMID 36254038

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the TUTOR study began on August 8, 2022, and 122 subjects were enrolled. Enrollment was completed on February 2, 2023. Per the protocol, a subject was considered enrolled once they had signed the informed consent form, met all inclusion and exclusion criteria, and completed carpal tunnel release (CTR) via their assigned treatment method.
Pre-assignment Details: No pre-assignments for this study
Groups:
- Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device: Participants who were randomized to and treated with the Carpal Tunnel Release with Ultrasound Guidance procedure using the UltraGuideCTR device in the TUTOR Study.
- Mini Open Carpal Tunnel Release (mOCTR): Participants who were randomized to and treated with the Mini Open Carpal Tunnel Release (mOCTR) procedure in the TUTOR Study.
Period: Overall Study
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Started | 94 | 28
Completed | 94 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mini Open Carpal Tunnel Release (mOCTR): Participants who were randomized to and treated using the Mini Open Carpal Tunnel Release (mOCTR) procedure in the TUTOR Study.
- Total: Total of all reporting groups
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR) | Total
Number analyzed (Participants) | 94 | 28 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 19 | 79
  >=65 years | 34 | 9 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 57 (14) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 21 | 81
  Male | 34 | 7 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 84 | 27 | 111
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 86 | 25 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ-SSS) Change
Description: The Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ-SSS) is a Carpal Tunnel Syndrome specific questionnaire that has been shown to be highly reproducible, internally consistent, valid, and responsive to clinical change in Carpal Tunnel Syndrome (CTS) and subject status post-carpal tunnel release (CTR). The BCTQ consists of 11 symptom severity questions (BCTQ-SSS). Scoring for the BCTQ- SSS ranges from 1 to 5, with higher scores indicating more severe symptoms, and is calculated as the mean of each response. The mean change scores in BCTQ-SSS from baseline to the 3-month follow-up are reported for each study group. Negative change scores indicate decreased symptom severity and positive change scores indicate increased symptom severity.
Time Frame: 3 Month Follow-Up
Population: Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ-SSS) change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 89 | 28
units on a scale | -1.5 [-1.6 to -1.4] | -1.5 [-1.7 to -1.4]
Statistical Analysis 1: Comparison: Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device vs Mini Open Carpal Tunnel Release (mOCTR); Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.13 to 0.29]

2. Primary Outcome: Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ-FSS) Change
Description: The Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ-FSS) additionally consists of 8 functional status questions. Scoring for the BCTQ-FSS ranges from 1 to 5, with higher scores indicating more functional limitation, and is calculated as the mean of each response. The mean change scores in BCTQ-FSS from baseline to the 3-month follow-up are reported for each study group. Negative change scores indicate decreased functional limitation and positive change scores indicate increased functional limitation.
Time Frame: 3 Month Follow-Up
Population: Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ-FSS) change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 89 | 28
units on a scale | -0.8 [-0.9 to -0.7] | -0.8 [-1.0 to -0.7]
Statistical Analysis 1: Comparison: Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device vs Mini Open Carpal Tunnel Release (mOCTR); Test type: Superiority; p = 0.92, Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.2 to 0.23]

3. Other Pre Specified Outcome: Participants With Device or Procedure Related Adverse Events
Description: Participants with adverse events (AEs) occurring within 90 days of treatment and that are adjudicated as definitely related or probably related to the device or definitely related or probably related to the procedure will be included in this endpoint. The incidence of device- or procedure-related AEs within 90 days of treatment in each study group will represent an endpoint of the study.
Time Frame: 3 Month Follow-Up
Population: Participants with Procedure and/or Device-Related Adjudicated Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 94 | 28
Participants | 2 | 1

4. Other Pre Specified Outcome: Numeric Pain Scale Change
Description: The Numeric Pain Scale measures pain severity. Scoring for the Numeric Pain Scale ranges from 0 (indicating no pain) to 10 (indicating worst pain possible). The mean change scores in the Numeric Pain Scale from baseline to the 3-month follow-up are reported for each study group. Negative change scores indicate decreased pain severity and positive change scores indicate increased pain severity.
Time Frame: 3 Month Follow-Up
Population: Numeric Pain Scale change at 3 months
Measure: Mean (95% Confidence Interval); unit: Unit
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 89 | 28
Unit | -3.2 [-3.5 to -2.8] | -3.8 [-4.4 to -3.2]
Statistical Analysis 1: Comparison: Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device vs Mini Open Carpal Tunnel Release (mOCTR); Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Net) = 0.61, 95% CI 2-sided [-0.08 to 1.3]

5. Other Pre Specified Outcome: EuroQol 5-Dimension 5-Level (EQ-5D-5L) Change
Description: The EuroQol 5-Dimension 5-Level (EQ-5D-5L) is a generic preference-based questionnaire developed by the EuroQol Group to measure health-related quality of life. The EQ-5D-5L measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking consisting of: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Scoring for the EQ-5D-5L ranges from -0.57 (indicating lowest quality of life) to 1.00 (indicating highest quality of life). The mean change scores in the EQ-5D-5L from baseline to the 3-month follow-up are reported for each study group. Negative change scores indicate decreased quality of life and positive change scores indicate increased quality of life.
Time Frame: 3 Month Follow-Up
Population: EuroQol 5-Dimension 5-Level (EQ-5D-5L) change at 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 89 | 28
units on a scale | 0.11 [0.09 to 0.14] | 0.12 [0.07 to 0.16]
Statistical Analysis 1: Comparison: Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device vs Mini Open Carpal Tunnel Release (mOCTR); Test type: Superiority; p = 0.9, Mixed Models Analysis; Mean Difference (Net) = 0, 95% CI 2-sided [-0.06 to 0.05]

6. Other Pre Specified Outcome: Time to Return to Work Among Employed Subjects
Description: The time to return to work will be defined as the number of days between treatment and the time the subject reports returning to work in any capacity.
Time Frame: 3 Month Follow-Up
Population: Time to return to work in days among employed subjects
Measure: Median (Full Range); unit: Days
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 56 | 19
Days | 3.0 [1.0 to 8.5] | 4.0 [1.0 to 15.0]

7. Other Pre Specified Outcome: Participants Who Returned to Normal Daily Activities Within 3 Days Postoperatively
Description: The time to return to normal daily activities will be defined as the number of days between treatment and the time the subject reports returning to normal daily activities, irrespective of work status.
Time Frame: 3 Month Follow-Up
Population: Participants who returned to normal daily activities within 3 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
Number analyzed (Participants) | 94 | 28
Participants | 55 | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected out to 1 year.
Description: AE could be reported 3 ways. 1) Documented by the site during the study procedure. 2) Subject reported an AE directly to the investigative site. 3) AE identified by the site during the review of the subject-uploaded wound healing images. If the site identifies a potential AE based on an image review or is notified of a potential AE by the subject, confirmation of the AE will occurred by phone call with the subject or by asking the subject to return for a follow-up clinical evaluation.
Arm/Group | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device | Mini Open Carpal Tunnel Release (mOCTR)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/28
Other Adverse Events (participants affected / at risk) | 1/94 | 1/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device (N=94) | Mini Open Carpal Tunnel Release (mOCTR) (N=28)
Nerve Injury - Digital-Median (Surgical and medical procedures) | 1 (1) | 0 (0) — Epineurial laceration without axonal disruption on the dorsal aspect of the third common digital nerve, 2 cm distal to its median nerve origin. A nerve wrap was placed and the incision was closed with sutures.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carpal Tunnel Release With Ultrasound Guidance Using the UltraGuideCTR Device (N=94) | Mini Open Carpal Tunnel Release (mOCTR) (N=28)
Nerve Injury - Digital-Median: Neurapraxia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Wound Dehiscence/ delayed healing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05405218/Prot_SAP_001.pdf